CLINICAL TRIAL: NCT02862600
Title: A Phase 2, Multi-Center, Open-Label, Ascending Dose Study on the Efficacy, Safety and Tolerability of Perhexiline in Patients With Hypertrophic Cardiomyopathy and Moderate to Severe Heart Failure With Preserved Left Ventricular Function
Brief Title: Open-Label Study of Perhexiline in Patients With Hypertrophic Cardiomyopathy and Moderate to Severe Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Heart Metabolics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HML-PHX-005
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Cardiomyopathy, Hypertrophic; Cardiomyopathy, Hypertrophic, Familial
Keywords: hypertrophic cardiomyopathy; heart failure; cardiopulmonary exercise testing; 6 minute walk test; perhexiline; carnitine palmitoyltransferase; mixed ion channel effects; late sodium current inhibitor; calcium channel inhibition
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathy, Hypertrophic, Familial; Heart Failure | interventions — Perhexiline

STUDY DESIGN:
Intervention Model Description: Open-label, 2 period, dose escalation study of perhexiline in symptomatic patients with hypertrophic cardiomyopathy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Perhexiline (Experimental): Perhexiline will be administered orally. Dosing will be determined based on plasma level monitoring. For the first 8 week period, the target range will be 100-300 ng/mL, for the second 8 week period, the target range will be 300-500 ng/mL.
  Interventions: Drug: Perhexiline; Device: Use of bioanalytical assay to monitor plasma levels of perhexiline

INTERVENTIONS:
Drug: Perhexiline — Period 1 (Weeks 1-8) and Period 2 (Weeks 9-16): dose titrated to two different plasma levels of perhexiline
Device: Use of bioanalytical assay to monitor plasma levels of perhexiline — The bioanalytical assay is the device under investigation. It will be used to monitor plasma levels of perhexiline. The data obtained from this analysis will be used to guide dose adjustments of perhexiline.

SUMMARY:
The purpose of this study is to evaluate the effect of perhexiline on exercise performance (efficacy) and safety in patients with hypertrophic cardiomyopathy and moderate-to-severe heart failure following dosing for 16 weeks.

DETAILED DESCRIPTION:
Patients with hypertrophic cardiomyopathy and symptoms without severe outflow obstruction will be eligible to participate. Enrollment will be limited to subjects who are unable to attain 75% of their maximum predicted MVO2 at cardiopulmonary exercise testing. Subjects with genetic evidence of CYP2D6 poor metabolizer status will be excluded.

Subjects will undergo functional testing at baseline with CPEX testing and 6 minute walk distance testing. They will begin perhexiline orally, and the dose will be adjusted according to plasma level testing. For the first 8 week period, the target therapeutic range will be 100-300 ng/mL, and for the second 8 week period, the range will be 300-500 ng/mL. Functional testing will be repeated at the end of both periods.

ELIGIBILITY:
Key Inclusion Criteria:

* Hypertrophic cardiomyopathy with symptoms of moderate-to-severe heart failure
* Left ventricular hypertrophy with maximum LV wall thickness ≥ 15 mm
* Left ventricular ejection fraction ≥ 50%
* Able to perform exercise testing but unable to exceed 75% of the predicted age-adjusted maximum level

Key Exclusion Criteria:

* CYP2D6 Poor Metabolizer (PM) status
* History of a known chronic liver disease
* ALT, AST, alkaline phosphatase, or LDH > 1.5 x upper limit of normal
* Total Bilirubin > 2.0 x upper limit of normal
* Severe LV outflow obstruction
* Asymptomatic patients or cardiomyopathy-related criteria as per protocol
* QT interval related criteria as per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Midei, MD, Study Chair — Heart Metabolics
Locations (11):
- United States (11):
  - Stanford, California
  - Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Detroit, Michigan
  - Columbus, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Germantown, Tennessee
  - Salt Lake City, Utah
  - Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty subjects were screened at 13 US centers. Of these, 36 were found suitable for enrollment, and 35 were enrolled prior to study termination.
Pre-assignment Details: The principal reason for screen failure was attainment of > 75% of the maximum predicted MVO2 on CPEX testing. One subject was found to be a CYP2D6 poor metabolizer.
Period: Period 1--Perhexiline-low Target Range
Arm/Group | Perhexiline
Started (Target range 100-300 ng/mL) | 35 (First subject underwent baseline functional assessment and perhexiline dosing on August 22, 2016)
Completed (Period and study terminated) | 22 (Study terminated on April 26, 2017 due to lack of efficacy.)
Not Completed | 13
Not completed — Lack of Efficacy | 9
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 1
Period: Period 2--Perhexiline-high Target Range
Arm/Group | Perhexiline
Started (Target range 300-500 ng/mL) | 22 (First subject completed Period 1 and moved into Period 2 perhexiline dosing on October 17, 2016)
Completed (Period and study termination) | 15 (Study terminated on April 26, 2017 due to lack of efficacy in first 15 subjects completing Period 2.)
Not Completed | 7
Not completed — Lack of Efficacy | 7

BASELINE CHARACTERISTICS:
Population: Baseline data was collected on all enrolled subjects on Day 0.
Arm/Group | Perhexiline
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 50 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of VO2MAX at 16 Weeks
Description: At the conclusion of 16 weeks of perhexiline treatment, MVO2 was measured using CPEX and compared to MVO2 measured at baseline.
Time Frame: end of Period 2 (Week 16)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Perhexiline--16 Weeks: Subjects completing 8 weeks of perhexiline at target range 100-300 ng/ml, and an additional 8 weeks of perhexiline at target range 300-500 ng/ml.
Arm/Group | Perhexiline--16 Weeks
Number analyzed (Participants) | 15
ml/kg/min | -0.2 (2.7)

2. Secondary Outcome: Change From Baseline of VO2MAX at End of Period 1
Description: At the conclusion of 8 weeks of perhexiline treatment, MVO2 was measured using CPEX and compared to MVO2 measured at baseline.
Time Frame: end of Period 1 (Week 8)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Perhexiline--8 Weeks: Subjects completing 8 weeks of perhexiline at target range 100-300 ng/ml.
Arm/Group | Perhexiline--8 Weeks
Number analyzed (Participants) | 22
ml/kg/min | 0.3 (1.8)

3. Secondary Outcome: Change From Baseline in the Six-minute Walk Test at the End of Period 2
Description: At the conclusion of 16 weeks of perhexiline treatment, 6MWD was measured and compared to 6MWD measured at baseline.
Time Frame: end of Period 2 (Week 16)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Perhexiline--16 Weeks
Number analyzed (Participants) | 15
meters | 27 (46)

4. Secondary Outcome: Change From Baseline in the Six-minute Walk Test at the End of Period 1
Description: At the conclusion of 8 weeks of perhexiline treatment, 6MWD was measured and compared to 6MWD measured at baseline.
Time Frame: end of Period 1 (Week 8)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Perhexiline--8 Weeks
Number analyzed (Participants) | 22
meters | 16 (50)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment (Day 0) until 30 days after study drug termination.
Groups:
- Perhexiline: All enrolled subjects
Arm/Group | Perhexiline
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 5/35
Other Adverse Events (participants affected / at risk) | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perhexiline (N=35)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1
Exacerbation of congestive heart failure (Cardiac disorders) | 1 — The subject had a history of CHF which was exacerbated during the study. The investigator classified the event as unrelated to study drug.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
atrial fibrillation recurrence (Cardiac disorders) | 1 — A subject with a history of AF had a recurrent event during the trial. The subject was admitted and the condition resolved. The investigator classified the event as unrelated to study drug.
recurrence of atrial fibrillation (Cardiac disorders) | 1 — A subject with a history of AF had a recurrent event during the trial. The subject was admitted and the condition resolved. The investigator classified the event as unrelated to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perhexiline (N=35)
Fatigue (General disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Influenza like illness (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2

LIMITATIONS AND CAVEATS:
Early termination due to lack of efficacy in the first 15 subjects completing the study. Any conclusions regarding safety or efficacy a challenging in light of the small numbers of subjects studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-12-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT02862600/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT02862600/SAP_001.pdf
  • Informed Consent Form (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT02862600/ICF_002.pdf